CLINICAL TRIAL: NCT03708887
Title: Double-blind and Placebo-controlled Study on Intervention Effect of n-3 Fatty Acids on Glucose and Lipid Homeostasis Disorders in Obese/Diabetic Populations
Brief Title: The Effect of Omega-3 FA on Glucose and Lipid Homeostasis Disorders in Obese/Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT-N3
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Hyperglycaemia (Diabetic); Hyperlipidemias
Keywords: Type 2 diabetes; Obesity; Omega-3 fatty acids
MeSH Terms: conditions — Hyperglycemia; Hyperlipidemias; Diabetes Mellitus, Type 2; Obesity | interventions — Drug and Narcotic Control

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): Low-dose omega-3 fatty acid supplementation, omega-3 fatty acids capsules, 1.5 grams per day for 1 year.
  Interventions: Drug: Low dose omega-3 fatty acid supplementation
- High dose group (Experimental): High-dose omega-3 fatty acid supplementation, omega-3 fatty acids capsules, 3 grams per day for 1 year.
  Interventions: Drug: High dose omega-3 fatty acid supplementation
- Control group (Placebo Comparator): Control drug, matching placebo capsules, 3 grams per day for 1 year.
  Interventions: Drug: Control drug

INTERVENTIONS:
Drug: Low dose omega-3 fatty acid supplementation — Omega-3 fatty acids capsules, 1.5 g/d by mouth for 1 year
  Other Names: Fish oil supplement
  Arms: Low dose group
Drug: High dose omega-3 fatty acid supplementation — Omega-3 fatty acids capsules, 3 g/d by mouth for 1 year
  Other Names: Fish oil supplement
  Arms: High dose group
Drug: Control drug — Matching placebo capsules,3 g/d by mouth for 1 year
  Other Names: Placebo drug
  Arms: Control group

SUMMARY:
A double-blind and placebo-controlled study is conducted in the current human study.

The purpose of this study is to investigate the effects of n-3 PUFA intervention on glucose and lipid homeostasis in Chinese diabetic/obese patients.

DETAILED DESCRIPTION:
Approximately 450 diabetic and 450 obese patients will be enrolled from Lanxi in China. They will be randomly assigned into one of the following three groups: Omega-3 fatty acids capsules (1.5 g/d); or omega-3 fatty acids capsules (3 g/d); or placebo capsules. Blood, feces and urine samples will be collected before and after treatment. Glucose and lipid parameters will be measured. Diabetes comorbidities and complications will also be assessed. This study will also explore the new mechanisms of n-3 PUFAs on improving glucose and lipid homeostasis and other outcomes based on multi-omics and establish a model for precision intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetes for diabetic groups according to WHO diagnostic criteria;
* BMI≥28 for obese groups;
* Aged between 40 and 75 years.

Exclusion Criteria:

* Type 1 diabetes;
* Cardiovascular disease;
* Cancer;
* Liver or kidney disease;
* Premenopausal women, pregnancy or lactation;
* Allergy to fish;
* Have participated in other clinical trials in the last three months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose from baseline | 12 months
  The investigators will measure HbA1c and fasting plasma glucose levels in blood samples before and after treatment.
Change in blood lipids from baseline | 12 months
  The investigators will measure Triglycerides (TG), total cholesterol (TC), LDL-C, and HDL-C levels in blood samples before and after treatment.
Change in carotid plaque and carotid intima-meida thickness | 12 months
  A FUJIFILM SonoSite ultrasound system will be used to assess carotid artery plaque lesions and measure carotid intima-media thickness (CIMT).

SECONDARY OUTCOMES:
Change in gut microbiota from baseline | 12 months
  The investigators will collect faeces sample from every participants and 16S rDNA sequencing will be used to analyze the composition of gut microbiota.
Change in sleep quality | 12 months
  The investigators will measure the Pittsburgh Sleep Quality Index (PSQI) through face-to-face questionnaire before and after treatment. The PSQI ranges from 0 to 21, with a higher score indicating a worse sleep quality.
Change in cognitive function | 12 months
  The investigators will do the mini-mental state examination (MMSE) before and after treatment. The MMSE score ranges from 0 to 30, with higher scores indicative of superior cognitive functioning.
Change in bone mineral density (BMD) | 12 months
  The whole body of the patient will be scanned and analyzed by a whole-body dual-energy X-ray absorptiometry (DXA) to measure the bone mineral density (BMD).
Change in body fat distribution | 12 months
  The whole body of the patient will be scanned and analyzed by a whole-body dual-energy X-ray absorptiometry (DXA) to measure the total and regional body fat mass (FM) and then percentages of regional body fat will be calculated.
Change in urinary protein concentration | 12 months
  The investigators will collect urine sample from every participant and measure urinary protein before and after treatment.
Change in estimated glomerular filtration rate (eGFR) | 12 months
  The investigators will collect blood sample from every participant and measure blood creatinine before and after treatment. The Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation will be used to calculate the eGFR.
Change in blood metabolome | 12 months
  The investigators will collect blood samples from every participant and the UPLC-MS/MS method will be used to analyze the blood metabolomics profile.

OTHER OUTCOMES:
Change in fecal metabolome | 12 months
  The investigators will collect fecal samples from every participant and the UPLC-MS/MS method will be used to analyze the fecal metabolomics profile.
Change in urine metabolome | 12 months
  The investigators will collect urine samples from every participant and the UPLC-MS/MS method will be used to analyze the urine metabolomics profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanxi Red Cross Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhuang P, Liu X, Jia W, Zheng W, Wan X, Chen W, Gu J, Li Y, Lan X, Li H, Tong W, Wu Y, Wu X, Ao Y, Ye H, Wu F, Zhu L, Zhang L, Li Y, Meng D, Tian Y, Wang A, Wu S, Zhu F, Zhang Y, Shi H, Yu X, Zhang F, Zhang Y, Jiao J. Marine n-3 fatty acid treatment for carotid plaques in patients with type 2 diabetes. Cardiovasc Diabetol. 2026 Jan 20. doi: 10.1186/s12933-026-03082-7. Online ahead of print. PMID 41559698
- [Derived] Zhuang P, Wu Y, Yao J, Liu X, Liu H, Wan X, Jia W, Wang T, Zhang Y, Jiao J. Marine n-3 polyunsaturated fatty acids slow sleep impairment progression by regulating central circadian rhythms in type 2 diabetes. Cell Rep Med. 2025 May 20;6(5):102128. doi: 10.1016/j.xcrm.2025.102128. Epub 2025 May 9. PMID 40347940